CLINICAL TRIAL: NCT05525065
Title: Investigating the Nature and Prevalence of Glucocorticoid-related Morbidity in Patients With Autoimmune Bullous Disease (AIBD) Using the Glucocorticoid Toxicity Index (GTI)
Brief Title: Investigating the Morbidity of Glucocorticoid Use in Patients With Autoimmune Bullous Diseases (AIBDs)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Premier Specialists, Australia (Other)
Collaborators: Steritas (Unknown)
Responsible Party: Sponsor
Other Study IDs: ABDF-GTI2021
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Autoimmune Bullous Dermatosis; Glucocorticoids Toxicity
MeSH Terms: interventions — Glucocorticoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with autoimmune bullous disease receiving glucocorticoids for the duration of the study: Patients with autoimmune bullous disease currently receiving glucocorticoids for their condition, as independently assessed by an appropriately qualified medical professional/dermatologist, for the duration of the study period.
  Interventions: Drug: GlucoCorticoid
- Patients with autoimmune bullous disease not currently receiving glucocorticoids: Patients with autoimmune bullous disease who have received glucocorticoids for their condition in the past, but are not currently on steroids.
- Patients with autoimmune bullous disease ceasing glucocorticoids during the study period: Patients with autoimmune bullous disease who initially had glucocorticoid treatment at the first visit, and had ceased glucocorticoid use during the study period.
  Interventions: Drug: GlucoCorticoid

INTERVENTIONS:
Drug: GlucoCorticoid — Glucocorticoid as calculated in prednisone oral equivalents.
  Groups: Patients with autoimmune bullous disease ceasing glucocorticoids during the study period; Patients with autoimmune bullous disease receiving glucocorticoids for the duration of the study

SUMMARY:
This project utilised the validated glucocorticoid toxicity index (GTI) tool to assess the morbidity of glucocorticoid-use in patients with autoimmune bullous disease. In particular, the study investigated the nature and prevalence of glucocorticoid-induced myopathy.

DETAILED DESCRIPTION:
This study is an multi-centre observational trial. Patients with AIBDs are recruited based on the criteria: an age of eighteen years or above; a new or established diagnosis of autoimmune bullous disease confirmed by clinical assessment, histopathology, immunofluorescence, and enzyme-linked immunoassay (ELISA) or biochip testing; new or current use of oral glucocorticoids for the treatment of autoimmune bullous disease (Group 1, active treatment group), patients with receipt of previous oral glucocorticoid use with no current use (Group 2, steroid-sparing control group) or patients who had ceased glucocorticoids during the study (Group 3, ceased steroid group) ; attendance of at least one baseline visit (V1) and one follow-up visit during the study period; and, the provision of capacitated and informed consent.

Patients are considered for enrolment based on inclusion criteria after attendance at a bullous disease clinic at a participating study site. At the baseline visit (V1), patients are comprehensively interviewed for demographic factors (age, gender), pre-existing medical conditions, and past and current medications. Patients attend regular follow-up visits at three-month intervals, to a maximum follow-up period of 15 months (V6). Treatment plans, including glucocorticoid dose, are determined by accredited medical professionals based on the clinical condition of the patient.

The Glucocorticoid Toxicity Index (GTI) tool (Figure 1) is used to evaluate glucocorticoid toxicity at all visits, including in dermatologic, neuropsychiatric, musculoskeletal, endocrine and metabolic domains.

Myopathy was measured and graded in accordance to the GTI.

Patients were divided into three groups: Group 1 (control) comprised of patients was comprised of who were not exposed to glucocorticoids during the study period, Group 2 comprised of patients whose glucocorticoid dose was ceased during the study period. Patients who continued on glucocorticoid treatment for the duration of the study period formed the third group.

ELIGIBILITY:
Inclusion Criteria:

* An age of eighteen years or above.
* A new or established diagnosis of autoimmune bullous disease confirmed by clinical assessment, histopathology, immunofluorescence, and enzyme-linked immunoassay (ELISA) or biochip testing
* New or current use of oral glucocorticoids for the treatment of autoimmune bullous disease (Group 1, active treatment group), or patients with receipt of previous oral glucocorticoid use with no current use (Group 2, steroid-sparing control group)
* Attendance of at least one baseline visit (V1) and one follow-up visit during the study period; and, the provision of capacitated and informed consent.

Exclusion Criteria:

* Inability to consent.
* Under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with autoimmune bullous disease who regularly attend a bullous clinic as part of their regular care. Patients who have either used glucocorticoids in the past or are currently using glucocorticoids.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Glucocorticoid Toxicity Score | 2 years
  Glucocorticoid toxicity score as calculated by the glucocorticoid toxicity index (GTI) application licenced by Steritas.
  The final glucocorticoid toxicity index (GTI) score is comprised of two sub-scores. The GTI-cumulative worsening score (GTI-CWS) captures any additive glucocorticoid toxicities, transient or persistent, that are not present at baseline is scored from 0 to +439. The GTI-aggregate improvement score (GTI-AIS) assesses end-point toxicity comparative to baseline and is scored from -317 to +410; a negative score represents an improvement in toxicity, whilst a positive score indicates worsening toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Dedee Murrell, MBBS, Study Chair — University of New South Wales
Locations (1):
- Premier Specialists, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No